CLINICAL TRIAL: NCT06421818
Title: Formula-to-Syndrome Effect and Pharmacomicrobiomics Mechanism of Colon Delivery of Baitouweng Decoction for Treating Large Intestine Damp-heat Syndrome of Ulcerative Colitis
Brief Title: Effect and Mechanism of Baitouweng Decoction for Large Intestine Damp-heat Syndrome of Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Faming Zhang, chief physician, PhD, The Second Hospital of Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTW-RCT
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Ulcerative Colitis
Keywords: Baitouweng Decoction; Formula-to-Syndrome Effect; Ulcerative colitis; Pharmacomicrobiomics; Colon delivery
MeSH Terms: conditions — Colitis, Ulcerative | interventions — baitouweng tang

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For groups receiving Baitouweng Decoction by oral administration and rectal edema，the interventions are single-blind to investigators and outcomes assessor. For groups receiving Baitouweng Decoction or placebo by colonic TET, the interventions are double-blind to participants, care provider, investigators and outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Colonic TET treatment group (Experimental): Baitouweng Decoction is administered through the colonic TET.
  Interventions: Drug: Baitouweng Tang
- Colonic TET placebo group (Placebo Comparator): The same volume of placebo as the colonic TET treatment group was administered through the colonic TET.
  Interventions: Other: Placebo
- Rectal enema group (Active Comparator): Baitouweng Decoction is administered through rectal enema.
  Interventions: Drug: Baitouweng Tang
- Oral group (Active Comparator): Baitouweng Decoction is administered through oral.
  Interventions: Drug: Baitouweng Tang

INTERVENTIONS:
Drug: Baitouweng Tang — Baitouweng Decoction is composed of four herbs: Baitouweng, Rhizoma coptidis, Phellodendri huangbai and Qin Pi.
  Other Names: Baitouweng Decoction
  Arms: Colonic TET treatment group; Oral group; Rectal enema group
Other: Placebo — The same volume and color as Baitouweng Decoction.
  Arms: Colonic TET placebo group

SUMMARY:
Baitouweng Decoction is traditionally used to treat large intestine damp-heat syndrome of ulcerative colitis (UC) by oral administration and rectal enema.The project applicant's invention of transendoscopic entral tubing (TET) has been used in Baitouweng Decoction for the treatment of UC across the whole colon, however, the efficacy have not been reported and the underlying mechanism is still unclear. Compared with oral and rectal enema, Baitouweng Decoction by colon TET can improve the therapeutic effect by increasing the concentration of drugs in the whole colon, which need to be verified. This project will reveal the prescription effect and drug-microbiome interaction mechanism of whole colon repeated administration of Baitouweng Decoction in the treatment of UC through clinical randomized controlled studies, deep intestinal dynamic sampling, integrated analysis of multi-omics and TCM prescription metabolomics studies, and provide key scientific basis for the establishment of a new approach of whole colon repeated administration of TCM and a new strategy for the treatment of UC.

DETAILED DESCRIPTION:
A multi-center randomized controlled study will be conducted to compare the efficacy differences and multi-omics changes of colon TET, rectal enema and oral Baitouweng Decoction in the control of intestine damp-heat syndrome of UC. Moreover，a group of patients was designed to receive blank carrier solution through colon TET tube. After the study, the patients in this group were given compensation treatment of fecal microbiota transplantation as an ethical protection measure.The colonic TET will be implanted into the intestine and the whole colon will be covered with Baitouweng Decoction. The treatment period is 10 days. The primary outcome measure is the changes of fecal calprotectin before and after oral, colonic TET and rectal enema administration. And the secondary outcomes measure are the changes of disease condition, Mayo score and safety. Deep intestine fluid, stool, blood and urine samples were collected before and after treatment to study the changes of microbiomes, metabolomics and immunoomics. Identify the difference of the key material basis of Baitouweng Decoction and analyze its mechanism comprehensively. The key beneficial and harmful bacteria were identified by comprehensive analysis. A total of not less than 144 subjects are expected to be included and divided into colonic TET treatment group, colonic TET placebo group, rectal enema group, and oral group according to a ratio of 1:1:1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with ulcerative colitis;
2. The patients are in mild to moderate active stage with Mayo score of 3-8.
3. Patients with damp-heat syndrome of large intestine according to TCM syndrome differentiation: according to the expert consensus on integrated traditional Chinese and Western medicine diagnosis and treatment of UC, the main symptoms are diarrhea, mucopurulent and bloody stool, abdominal pain, and tenesmus. Secondary symptoms: anal burning, body heat is not Yang, dry mouth and bitter mouth, short red urine. Tongue pulse: tongue red fur yellow greasy, pulse slippery number. The determination of the above 8 syndromes can be made if there are 2 main symptoms and 1-2 secondary symptoms. The tongue pulse is for reference only.
4. The patients who can tolerate Baitouweng Decoction;
5. The patients who tolerance to colonoscopy and TET;
6. The patients who know and agree to participate in the clinical trial.

Exclusion Criteria:

1. The patients are complicated with other diseases that may cause diarrhea, such as infectious colitis, radiation enteritis, Crohn's disease, etc.
2. Patients with heart, brain, lung, liver, kidney and other serious diseases;
3. Patients do not cooperate to complete the clinical trial process;
4. Other cases considered unsuitable for inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The concentration of fecal calprotecin. | Baseline; Day 15; Day 53
  To compare the concentration of fecal calprotecin before and after oral, colonic TET and rectal enema administration.

SECONDARY OUTCOMES:
The change of Mayo score. | Baseline; Day 15; Day 22; Day 53; Day 99.
  To compare the change of Mayo score before and after oral, colonic TET and rectal enema administration. The Mayo score included the number of bowel movements, blood in the stool, endoscopic findings and overall physician evaluation. The total score was 12 points. The higher the score, the higher the degree of disease activity.
Incidence of Treatment-Emergent Adverse Events | Day 15; Day 22; Day 53; Day 99.
  The number of adverse reactions that are associated with Baitouweng Decoction reported by subjects from the start of treatment to the end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Department of Microbiota Medicine & Medical Centre for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang W, Lu G, Wu X, Wen Q, Zhang F. Colonic Transendoscopic Enteral Tubing Is a New Pathway to Microbial Therapy, Colonic Drainage, and Host-Microbiota Interaction Research. J Clin Med. 2023 Jan 18;12(3):780. doi: 10.3390/jcm12030780. PMID 36769429
- [Result] Zhang X, Zhang L, Chan JCP, Wang X, Zhao C, Xu Y, Xiong W, Chung WC, Liang F, Wang X, Miao J, Bian Z. Chinese herbal medicines in the treatment of ulcerative colitis: a review. Chin Med. 2022 Apr 4;17(1):43. doi: 10.1186/s13020-022-00591-x. PMID 35379276
- [Result] Gou H, Su H, Liu D, Wong CC, Shang H, Fang Y, Zeng X, Chen H, Li Y, Huang Z, Fan M, Wei C, Wang X, Zhang X, Li X, Yu J. Traditional Medicine Pien Tze Huang Suppresses Colorectal Tumorigenesis Through Restoring Gut Microbiota and Metabolites. Gastroenterology. 2023 Dec;165(6):1404-1419. doi: 10.1053/j.gastro.2023.08.052. Epub 2023 Sep 12. PMID 37704113
- [Result] Wei P, He Q, Liu T, Zhang J, Shi K, Zhang J, Liu S. Baitouweng decoction alleviates dextran sulfate sodium-induced ulcerative colitis by suppressing leucine-related mTORC1 signaling and reducing oxidative stress. J Ethnopharmacol. 2023 Mar 25;304:116095. doi: 10.1016/j.jep.2022.116095. Epub 2022 Dec 26. PMID 36581160
- [Result] Gu X, Miao Z, Wang Y, Yang Y, Yang T, Xu Y. New Baitouweng decoction combined with fecal microbiota transplantation alleviates DSS-induced colitis in rats by regulating gut microbiota metabolic homeostasis and the STAT3/NF-kappaB signaling pathway. BMC Complement Med Ther. 2022 Nov 24;22(1):307. doi: 10.1186/s12906-022-03766-z. PMID 36424592